CLINICAL TRIAL: NCT06165237
Title: A Phase I Clinical Trial to Evaluate the Drug-drug Interaction and Safety Between "BR6001-1" and "BR6001-2" in Healthy Adult Volunteers
Brief Title: A Study to Evaluate the Drug-drug Interaction and Safety Between "BR6001-1" and "BR6001-2"
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BR-ARC-CT-101
Record Dates: First submitted 2023-12-03; First posted 2023-12-11 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Gastric or Duodenal Ulcer
MeSH Terms: conditions — Duodenal Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BR6001-1+BR6001-2 (Experimental)
  Interventions: Drug: BR6001-1; Drug: BR6001-2

INTERVENTIONS:
Drug: BR6001-1 — One tablet administered alone, Once a day
Drug: BR6001-2 — One tablet administered alone, Once a day

SUMMARY:
The purpose of this clinical trial is to evaluate the drug-drug interaction and safety between "BR6001-1" and "BR6001-2" in healthy adult volunteers

ELIGIBILITY:
Inclusion Criteria:

* Those who weigh 50 kg or more and have body mass index (BMI) within the range of 18.0 to 30.0kg/m² at screening visit.
* Those who sign written consent spontaneously to follow the study directions after listening to and understanding sufficient explanation of this clinical trial.

Exclusion Criteria:

* Those who have a medical history of gastrointestinal diseases(Crohn's disease, ulcer, acute or chronic pancreatitis, etc.) or gastrointestinal surgery (Except for simple appendectomy, hernia surgery) that may affect the absorption of investigational products.
* Those who have hypersensitivity reaction to investigational products or their additives in addition to other painkillers, anti-inflammatory drugs, antirheumatic drugs, benzimidazole.
* Those who have a history of clinically significant hypersensitivity reaction.
* Those taking anticoagulants, atazanavir, Rilpivirine and methotrexate.
* Those who eat an abnormal food that may affect the absorption, distribution, metabolism and excretion of investigational products or who eat food that may affect drug metabolism.
* Those who take any prescription drugs(including herbal medicines) that may affect characteristics of investigational product within 14 days prior to the date of first administration or who take any over-the-counter (OTC) drugs or vitamins within 10 days prior to the date of first administration (however, if it don't affect subject's safety and study's result according to the judgment of the investigator, they may participate in the study.)
* Those who take inducer and inhibitor of drug metabolizing enzymes such as barbiturates, etc. within 1 month prior to the first administration

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-03-30 (Actual); Primary Completion 2023-05-09 (Actual); Study Completion 2023-05-09 (Actual)

PRIMARY OUTCOMES:
AUCτ,ss | 0~24 hours after administration
  Area under the Plasma Concentration-Time Curve During Dosing Interval (tau) at Steady State
Cmax,ss | 0~24 hours after administration
  Maximum Concentration of Drug in Plasma at Steady State
The change(%) of Aspirin Reaction Units(ARU) & Thromboxane B2 (TxB2) at 24h after repeated administration (last administration date) compared to baseline (first administration date) | 0, 6, 24 hours after administration

CONTACTS AND LOCATIONS:
Locations (1):
- ChungBuk National University Hospital, Jungbuk, South Korea

IPD SHARING:
Plan to Share IPD: No